CLINICAL TRIAL: NCT02213757
Title: Effect of Vaginal Estrogen on Asymptomatic Microhematuria (AMH): A Randomized Controlled Trial [EVER Study]
Brief Title: Effect of Vaginal Estrogen on Asymptomatic Microhematuria (AMH)
Acronym: EVER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-071
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Microscopic Hematuria
Keywords: Hematuria; Menopause; Urinalysis
MeSH Terms: conditions — Hematuria

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premarin vaginal cream (Experimental): Premarin vaginal cream to be applied intra-vaginally and to vulva as follows: 1 gram nightly for 2 weeks, followed by 0.5 gram twice weekly for 6 weeks.
  Interventions: Drug: Premarin vaginal estrogen cream
- Placebo vaginal cream (Placebo Comparator): Placebo vaginal cream to be applied intra-vaginally and to vulva as follows: 1 gram nightly for 2 weeks, followed by 0.5 gram twice weekly for 6 weeks.
  Interventions: Drug: Placebo vaginal cream

INTERVENTIONS:
Drug: Premarin vaginal estrogen cream
  Other Names: Conjugated estrogens vaginal cream
  Arms: Premarin vaginal cream
Drug: Placebo vaginal cream — Inactive vaginal cream manufactured to mimic Premarin vaginal cream
  Other Names: Other names have not been specified
  Arms: Placebo vaginal cream

SUMMARY:
The purpose of this study is to determine if vaginal estrogen use is associated with resolution of blood in the urine (microscopic hematuria) in postmenopausal women. The hypothesis is that postmenopausal women with blood in the urine (microscopic hematuria) will have higher rates of resolution of hematuria after treatment course with vaginal conjugated equine estrogen cream compared to placebo cream

DETAILED DESCRIPTION:
This is a randomized controlled trial of vaginal estrogen cream for postmenopausal women with microscopic hematuria (AMH). Potential subjects will be screened with a dipstick urinalysis of a catheterized urine specimen, followed by microscopic urinalysis and urine culture if urine dipstick is positive for trace blood or greater. Women who are identified as having asymptomatic microscopic hematuria (>3 red blood cells (RBC) per high powered field (hpf)) on a single urine microscopy specimen in the absence of urinary tract infection or other benign cause will be eligible for enrollment.

Women meeting inclusion criteria will be randomized to either conjugated equine estrogen cream (Premarin, 0.625mg conjugated estrogens) or placebo cream for 8 weeks. Microscopic urinalysis of a catheterized urine specimen will be re-checked at 8 weeks to check for reduction, resolution or persistence of AMH. During the 8 weeks of vaginal estrogen or placebo, women will complete the recommended AMH workup as dictated by the American Urologic Association (AUA) guidelines (cystourethroscopy, serum blood urea nitrogen and creatinine levels, and computed tomography (CT) scan of the abdomen and pelvis with and without intravenous contrast).1

Validated questionnaires to assess vaginal atrophy and symptoms of urinary urgency and frequency will be completed at time of randomization and again at 8 weeks. Cost analysis of the standard AMH workup (cystourethroscopy and CT scan) versus empiric treatment with 8 weeks of vaginal estrogen cream will be calculated based on Medicare reimbursement, as well as market price for vaginal estrogen cream Additionally, patients will be asked to complete a questionnaire to assess the level of bother associated with completing the current AMH workup of CT scan and cystoscopy as compared to completing a treatment course of vaginal estrogen cream.

Secondary analyses will determine whether there are additional benefits to a trial period of vaginal estrogen cream in postmenopausal women with AMH prior to reflexively screening for urinary tract abnormalities. We will compare the cost of a standard AMH workup to a treatment course of vaginal estrogen cream, to determine whether vaginal estrogen with potential resolution of AMH is associated with any savings prior to pursuing further workup. Additionally, questionnaires will ask study participants whether they would prefer to undergo the current AUA AMH workup or a treatment course of vaginal cream, in order to assess bother and anxiety associated with these interventions.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women
* Asymptomatic microscopic hematuria (three or more red blood cells per high powered field on a single urine microscopy) in the absence of urinary tract infection.

Exclusion Criteria:

* Known urologic disease
* Presence of gross hematuria
* Presence of indwelling urologic foreign body (foley catheter, ureteral stent)
* Inability to obtain intravenous contrast CT scan (elevated creatinine, severe contrast allergy)
* History of pelvic irradiation or malignancy
* Not a candidate for vaginal estrogen

  * Allergy to vaginal estrogen
  * Current or prior diagnosis of breast or endometrial cancer
  * History of deep vein thrombosis/pulmonary embolus
  * Hypercoagulable state

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl B Iglesia, MD, Principal Investigator — Medstar Health Research Institute; Lee A Richter, MD, Study Director — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu JM, Williams KS, Hundley AF, Jannelli ML, Visco AG. Microscopic hematuria as a predictive factor for detecting bladder cancer at cystoscopy in women with irritative voiding symptoms. Am J Obstet Gynecol. 2006 May;194(5):1423-6. doi: 10.1016/j.ajog.2006.01.053. Epub 2006 Mar 30. PMID 16579943
- [Background] Shalom DF, Lin SN, St Louis S, Lind LR, Winkler HA. The prevalence of microscopic hematuria in women with pelvic organ prolapse. Female Pelvic Med Reconstr Surg. 2011 Nov;17(6):290-2. doi: 10.1097/SPV.0b013e3182357afb. PMID 22453223
- [Background] Jung H, Gleason JM, Loo RK, Patel HS, Slezak JM, Jacobsen SJ. Association of hematuria on microscopic urinalysis and risk of urinary tract cancer. J Urol. 2011 May;185(5):1698-703. doi: 10.1016/j.juro.2010.12.093. Epub 2011 Mar 21. PMID 21419446

RESULTS

PARTICIPANT FLOW:
Groups:
- Premarin Vaginal Cream: Premarin vaginal cream to be applied intra-vaginally and to vulva as follows: 1 gram nightly for 2 weeks, followed by 0.5 gram twice weekly for 6 weeks.
  Premarin vaginal estrogen cream
Period: Overall Study
Arm/Group | Premarin Vaginal Cream | Placebo Vaginal Cream
Started | 15 | 14
Completed | 10 | 10
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Premarin Vaginal Cream | Placebo Vaginal Cream | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 5 | 11
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resolution of Microscopic Hematuria
Description: Microscopic urinalysis will be performed after an 8 week trial of vaginal estrogen or placebo. Resolution of microscopic hematuria is defined according to AUA guidelines, <3 red blood cells per high powered field.
Time Frame: 8 weeks
Population: There were 14 participants in Placebo arm, 10 completed study and 4 were lost to follow up. 6 in Placebo group had resolution of microhematuria.
  There were 15 participants in Estrogen arm, 10 completed study and 5 were lost to follow up. 10 in Estrogen group had resolution of microhematuria.
Measure: Number; unit: participants
Arm/Group | Premarin Vaginal Cream | Placebo Vaginal Cream
Number analyzed (Participants) | 10 | 10
participants | 10 | 6

2. Secondary Outcome: Number of Participants With Improvement in Symptoms of Urinary Frequency and Urgency
Description: To determine the effect of vaginal estrogen compared to placebo on symptoms of urinary frequency and urgency. Participants that experience at least one point reduction in OAB-q score will qualify as a participant with improvement in these symptoms.
Time Frame: 8 weeks
Population: OAB-q scores were collected at baseline and at follow-up. Subjects with at least one point reduction in OAB-q score were recorded to show improvement in OAB-q score. Seven participants in the test group showed a reduction of at least 1 point and seven participants in the control group showed a reduction of at least 1 point.
Measure: Count of Participants; unit: Participants
Arm/Group | Premarin Vaginal Cream | Placebo Vaginal Cream
Number analyzed (Participants) | 10 | 10
Participants | 7 | 7

ADVERSE EVENTS:
Arm/Group | Premarin Vaginal Cream | Placebo Vaginal Cream
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No